CLINICAL TRIAL: NCT00263068
Title: An Open-Label Extension Trial to Investigate the Safety and Tolerability of Long-Term Treatment With Transdermal Rotigotine in Subjects With Idiopathic Restless Legs Syndrome
Brief Title: An Extension Trial to Investigate Long-Term Treatment With Transdermal Rotigotine in Idiopathic Restless Legs Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Study Director, UCB
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0793
Record Dates: First submitted 2005-12-05; First posted 2005-12-07 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Restless Legs Syndrome
Keywords: IDIOPATHIC RESTLESS LEGS SYNDROME
MeSH Terms: conditions — Restless Legs Syndrome | interventions — rotigotine

ARMS (1):
- 1 (Experimental): Up to 6.75 mg/day (optimal dosing)
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Drug: Rotigotine — Transdermal Patch 1 per day for 24 hours containing:
  1.125mg/day 2.25mg/day 4.5mg/day 6.75mg/day

SUMMARY:
This is a multicenter, open-label trial to assess safety and tolerability of rotigotine (SPM 936) in subjects with idiopathic Restless Legs Syndrome (RLS), administered at an optimal dose for up to 1 year. Subjects who successfully completed the Maintenance Period and the Taper Period of SP792 are allowed to enroll in this trial.

All subjects will begin the Titration Period at a daily dosage of 1.125mg rotigotine (2.5cm2 patch). Subjects will be up-titrated at 7-day intervals in 1.125mg (2.5cm2 increments, initial titration step only) and 2.25mg intervals (5cm2) increments to a maximum dose of 6.75mg/day (15cm2) rotigotine. The maximum length of titration is 28 days (±3 days), although not all subjects will require 28 days to reach their optimal dose.

A subject's dose may be increased or decreased, as needed by the investigator to maintain a subject's effective dose during the Maintenance Period. A Taper Period is provided to allow for safe, gradual withdrawal from trial medication

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic restless legs syndrome

Exclusion Criteria:

* Subject has an ongoing serious adverse event from SP792 that is assessed to be related to the trial medication by the investigator and/or the sponsor.
* Subject is pregnant, nursing, or is a woman of child-bearing potential who is not surgically sterile, 2 years postmenopausal, or does not consistently use 2 combined effective methods of contraception, including at least 1 barrier method, unless sexually abstinent.
* Subject has any medical or psychiatric condition that, in the opinion of the investigator, can jeopardize or would compromise the subject's ability to participate in this trial.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be assessed by adverse events, changes in laboratory tests, changes in vital signs, physical and neurological examination, changes in menstrual and sexual function, global subject rating | 1 year

SECONDARY OUTCOMES:
To obtain data on changes in severity in RLS symptoms and quality of life over a one year maintenance period. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- Schwarz, RTP, North Carolina, United States